CLINICAL TRIAL: NCT05521360
Title: Autonomic Modulation Training: A Biological Approach to Building Resilience and Wellness Capacity Among Police Exposed to Post-Traumatic Stress Injuries (PTSI)
Brief Title: Autonomic Modulation Training for Police Exposed to Post-Traumatic Stress Injuries
Acronym: AMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Judith Andersen, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CIHR Grant#433650; 39478 (Other: University of Toronto Research Ethics Board)
Record Dates: First submitted 2021-09-09; First posted 2022-08-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Stress, Physiological; Stress, Psychological
Keywords: Post Traumatic Stress Symptoms; Depressive Symptoms; Anxiety Symptoms; Operational Stress; Organizational Stress; Police; HRV Biofeedback; Psychophysiology
MeSH Terms: conditions — Stress, Psychological; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either the experimental or matched wait-list control group.
Who Masked: Outcomes Assessor
Masking Description: De-identified and masked data will be analyzed by an independent outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants randomized to the experimental group will complete baseline assessments, the 6 week AMT treatment online and then complete the follow up assessment (8 weeks total)
  Interventions: Behavioral: Autonomic Modulation Training
- Control (No Intervention): Participants randomized to the control group will be matched to the experimental group on demographic and outcome measures. Control participants will take the baseline assessments, will wait 7 weeks and take the follow-up assessment (8 weeks total). Control group participants are able to enrol in the AMT intervention at the end of their wait-list control period.

INTERVENTIONS:
Behavioral: Autonomic Modulation Training — AMT is a six week online behavioral intervention comprised of two components. The first component is an adapted (to online format) version of an established and publicly available HRVBF protocol (Lehrer et al, 2013, Biofeedback).The second is the integration of meta-cognitive coping skills and autonomic modulation breathing techniques into the HRVBF protocol (Arpaia & Andersen, 2019 Frontiers in Psychiatry; Andersen, Arpaia & Gustafsberg, 2021 Int J Emerg Ment Health and Human Resilience).
  Other Names: Heart Rate Variability Biofeedback (HRVBF) and Meta-Cognitive Skills for Post-traumatic Stress Injuries; AMT: Fitness for the Brain and Body
  Arms: Experimental

SUMMARY:
Police officers are exposed to hazardous, disturbing events that impose stress and long-term trauma. Upwards of 15-26% of public safety personnel (PSP) report one or more mental health symptoms. Accumulated stress and posttraumatic stress injuries (PTSI) result in chronic physical and mental health disorders including anxiety, depression, substance abuse, and cardiovascular disease. PTSI are related to reduced occupational performance, absenteeism, and risky behaviour, with implications for both police and public safety. Recent empirical evidence and government reports highlight a mental health and suicide crisis among various PSP sectors in Canada. Prior research forms an urgent call for evidence-based programs that build resilience and wellness capacity to prevent PTSI symptoms before they manifest as severe, chronic, diagnosable disorders. The current study addresses the limited effectiveness issues associated with existing interventions for PTSI among PSP and also considers sex and gender as central determinants of health.

Advances in physiology and neuroscience demonstrate that resilience is maintained by the healthy functioning of psychophysiological systems within the body. Objective biological measures have shown that chronic stress and trauma disrupt both psychological and physiological functioning, eroding resilience and reducing wellness capacity. Traditional interventions to build resilience among PSP have not adequately addressed the physiological underpinnings that lead to mental and physical health conditions, as well as burnout and fatigue following trauma. Together with previous empirical research lead by the NPA, the current proposal addresses this gap in PSP intervention research by employing Autonomic Modulation Training (AMT), a biological approach to building resilience and wellness capacity among PSP exposed to PTSI. Prior research shows that core AMT techniques effectively reduce psychophysiological stress and mental health symptoms in clinical and non-clinical populations. Further, research has shown that AMT techniques improve police health and occupational performance when completed during scenario-based, in-person training.

The aim of the proposed study is to test if a web-based delivery of AMT for police officers can build resilience and wellness capacity, and reduce symptoms of PTSI with similar effectiveness as in-person training. An additional novel scientific contribution of the current proposal includes an examination of sex and gender in baseline biological presentation of PTSI among police, and in response to a resilience building intervention.

DETAILED DESCRIPTION:
Hypotheses

Self-reported PTSI symptoms and resilience

H1. Symptoms of PTSI will be significantly reduced following completion of the AMT intervention, as measured by the Personal Health Questionnaire (PHQ-8), General Anxiety Disorder Scale (GAD-7), Depression, Anxiety, and Stress Scale (DASS), PTSD checklist (PCL-5), Copenhagen Burnout Inventory (CBI), Perceived Stress Scale (PSS), Alcohol Use Disorder Identification Test (AUDIT). Occupational/operational stress exposure will be measured by the Police Stress Questionnaire (PSQ) to account for possible exposures to stress and potentially traumatic events over the course of the intervention. Self-reported and COVID related stress will also be evaluated.

H2. Functional wellness capacity and resilience will be significantly improved following completion of the AMT intervention, as measured by the Brief COPE, Resilience Scale for Adults (RSA-33), and Brief Resilience Scale (BRS), White Bear Suppression Inventory (WBSI), Perseverative Thinking Questionnaire (PTQ), Ultra-Brief Penn State Worry Questionnaire (UB-PSWQ), Ultra-Brief Rumination Response Styles (UB-RRS), Good Health Practices Scale (GHPS).

H3. Sex and gender differences in PTSI will be observed at baseline and post-intervention assessment. We expect that females will report more symptoms of PTSI and lower resilience at baseline, and a greater reduction of PTSI symptoms and greater increase in resilience at follow-up than males. Gender role stress, discrimination, and harassment will be explored as moderators of PTSI symptoms at baseline and in response to the AMT intervention. Sex is measured by self-reported sex at birth, gender discrimination is measured by Workplace Gender Discrimination Scale (WGDS) and harassment is measured by the Gender Experiences Questionnaire (GEQ).

Objective biological indicators of PTSI symptoms and resilience

H4. Resting HRV will significantly increase following completion of the AMT intervention. Changes in resting HRV will be measured by time and frequency domain parameters based on data collected from the wearable HR monitors (e.g., high and low frequency HRV, LF/HF ratio, and the root mean square of successive differences (RMSSD) as recommended in the standards of practice for HRV analysis.

H5. RSA will significantly increase following completion of the AMT intervention. RSA is measured by obtaining the respiratory frequency. Greater power at the respiratory frequency indicates a higher level of RSA and will be analyzed using the gold standard HRV analysis program, Kubios.

H6. Recovery from acute stress will significantly improve following completion of the AMT intervention. Acute stress will be induced by completion of the online Paced Auditory Serial Addition Test (PASAT) and the Stroop Emotion Face Interference Task. Acute stress recovery will be assessed via a time domain measure of HRV (RMSSD).

H7. Based on inconsistencies in the extant literature, we will conduct exploratory analyses of any potential sex and gender differences in HRV, RSA, and acute stress recovery at baseline and post-intervention assessments. Although we expect to see improvements in self-reported and objective measures of PTSI and resilience overall (i.e., independent of sex and gender), we hypothesize that gender role stress and gender discrimination will moderate these effects. Further, it is possible that the magnitude of post-intervention changes is greater among women given the additional burden of exposure to a hyper-masculinized working environment. Because AMT provides tools for effective stress management, women may find more benefit from the intervention in managing the wider array of sociocultural stressors they experience compared to males.

ELIGIBILITY:
Inclusion Criteria:

* Current employment as an active duty (i.e., not on an extended medical or disability leave) frontline law enforcement officer in Canada.
* Must be fluent in English.

Exclusion Criteria:

* Non-Canadian law enforcement officers. Police administrators and civilian employees (i.e., non-sworn members) are not eligible.
* Officers that do not have weekly access to a personal computer to complete the online AMT intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic stress disorder (PTSD) symptoms | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  PTSD Checklist (PCL-5); a 20-item self-report measure of the 20 DSM5 PTSD symptoms experienced in the last month on a 5-point Likert scale ("Not at all" [0] - "Extremely" [4]). Total score range 0-80, with higher scores representing higher severity in PTSD symptoms, and provisional PTSD diagnosis cutoff at a score of 31 or higher.
Depression symptoms | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  Personal Health Questionnaire (PHQ-8): an 8-item self-report questionnaire for screening, diagnosing monitoring, and measuring depression severity over the last 2 weeks on a severity index ("Not at all" [0] - "Nearly Every day" [3]). Total score range 0-24, with a score of 10 or greater is considered major depression, 20 or more is severe major depression.
Global psychological symptoms | From baseline to follow-up (immediate post intervention assessment)
  Outcome measure:
  Depression, Anxiety, and Stress (DASS-42): a 42-item questionnaire where participants respond on a 4-point severity/frequency scale ("Did not apply to me at all" [0] - "Applied to me very much/most of the time" [3]) what degree they experienced each state over the last week. Total score range 0-42, with threshold cutoff for symptomatic depression, anxiety, or psychological distress at scores of 10, 8, 15 or greater for each subscale, respectively.
Anxiety symptoms | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  General Anxiety Disorder Scale (GAD-7): a 7-item self-report questionnaire measuring generalized anxiety disorder (GAD) symptoms on a severity index ("Not at all" [0] - "Nearly every day" [3]) experienced over the last 2 weeks. Total score range 0-21, with higher scores representing higher severity in GAD symptoms, and a cutoff score of 10 or greater for provisional cases of GAD.
Alcohol use | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  Alcohol Use Disorder Identification Test (AUDIT): a 10-item self-report measuring alcohol consumption, drinking behaviour, and alcohol related problems over the past year. Participants respond to questions on a 4-point scale ("Never" [0] - "Daily/Almost daily" [4]). Total score range 0-40, A score of 8 or more is associated with harmful or hazardous drinking, a score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence.
Perceived stress | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  Perceived Stress Scale (PSS): a 10-item self-report questionnaire measuring an individual's perceived life stress on a scale from ("Never" [0] - "Nearly every day" [3]) experienced over the last month. Total score range 0-40 with higher scores indicating higher perceived stress and cutoffs for low (0-13), moderate (14-26), and high (27-40) levels of stress.
Self-reported stress | From baseline to follow-up (immediate post intervention assessment) and session-to-session changes
  Global ratings of self-reported stress will be asked at the beginning of each AMT session using a sliding visual analog scale (VAS) ("Not at all stressful" [0] to "Extremely stressful" [10]) in response to two questions ('How stressful was this past week?' and 'How stressed are you right now?).
COVID stress experience | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  COVID adapted version of the Holmes Rahe Stress Inventory (HRSI): a list of 43 stressful life events that may contribute to illness. Each event has an assigned number of life change units, the sum of life change units creating the total score (range 0-1467). Higher scores indicate increased risk of stress-induced health breakdown from stress, with cutoffs for low susceptibility (<150), 50% chance (150-300), and 80% chance (300+) of a stress-induced health breakdown in the next 2 years.
Burnout symptoms | From baseline to follow-up (immediate post intervention assessment)
  Copenhagen Burnout Inventory (CBI)-personal burnout subscale: a 6-item self report questionnaire in which participants respond to experiences of prolonged physical and psychological exhaustion on a 5-point likert scale ("Never" [0]; "Seldom" [50]; Often [75]; "Always" [100]). Total score is the average of scores across the items (score range 0-100), with higher scores indicating higher levels of burnout.
Occupational police stress | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  Police Stress Questionnaire (PSQ): A 40-item self report questionnaire consisting of two subscales measuring job content (organizational stressors - 20 questions) and job context (operational stressors - 20 questions) on a 7-point Likert scale ("No stress" [1] - "Moderate stress" [4] - "A lot of stress" [7]) experienced over the last 6 months. Total score range for each subscale 20-140, with higher scores representing higher severity of stress experienced in the workplace.
Coping | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  Coping (Brief-COPE): a 28-item self report questionnaire measuring uses of different coping methods to a stressful event on a 4-point Likert scale ("I haven't been doing this at all" [1] - "I've been doing this a lot" [4]) across a number of coping style categories. The scale determines an individual's primary coping styles (total score range 28-72) with higher scores representing higher degree the individual engages in that coping style.
General resilience | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  Brief Resilience Scale (BRS); a 6-item self-report measuring general resilience and ability to cope with difficulty and stress on a 5-point Likert scale ("Strongly disagree" [1] - "Strongly agree" [5]). Index score equals average score response (range 1-5). Cutoffs for low (1-2.99) normal (3-4.3), and high (4.31-5) levels of resilience. Resilience scores are expected to increase following intervention.
Social resilience | From baseline to follow-up (immediate post intervention assessment)
  Outcome measure: Resilience Scale for Adults (RSA-33); a 33-item self-report scale measuring specific social protective factors presumed to enhance resilience among adults on a 5-point Likert Scale ("Strongly disagree" [1] - "Strongly agree" [5]). Factors including perception of self, planned future, social competence, social style, family cohesion, social resources. Mean scores are calculated for each subfactor. Increasing scores suggest higher levels of protective factors.
Thought suppression | From baseline to follow-up (immediate post intervention assessment)
  Outcome measure: The White Bear Suppression Inventory (WBSI) is a 15-item instrument that estimates thought processes on "suppression" and "intrusion" dimensions based on a 5-point Likert scale ("Strongly disagree" [1], "Strongly agree" [5]). Scores range from 15 to 75, with higher scores indicating a greater tendency to suppress thoughts.
Repetitive thinking | From baseline to follow-up (immediate post intervention assessment)
  Outcome measure:
  Perseverative Thinking Questionnaire (PTQ): 15 items assessing repetitive negative thinking (RNT) using a 5-point Likert scale from ("Never" [0] - "Almost Always" [4]). A higher score (total range 0-60) on reflects a high level of RNT.
Worry | From baseline to follow-up (immediate post intervention assessment)
  Outcome measure: Ultra Brief-Penn State Worry Questionnaire (UB-PSWQ): 16 items that measure a trait-like tendency to worry, focusing on the dimensions of frequency, controllability, and distress on a Likert-scale ("Not at all typical of me" [1] - "Very typical of me" [5]); total score range 16-80, higher scores indicate higher levels of worry.
Rumination | From baseline to follow-up (immediate post intervention assessment)
  Outcome measure: Ultra-Brief Rumination Response Styles (UB-RRS) Questionnaire: 5 item self-report questionnaire on rumination frequency when depressed on a 4-point Likert scale ("Almost Never" [1] - " Almost Always" [4]); total score range 5-20, with higher scores indicating higher degrees of ruminative symptoms.
Good health practices | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  Good Health Practices Scale (GHPS): a 16-item self-report scale of health behaviour statements (ex. I exercise to stay healthy, I eat a balanced diet, I see a dentist for regular checkups) on a 5-point Likert scale ("Not at all like me" [1] - "Very much like me" [5]). Total score range 16-80, with higher scores representing higher amounts of good health practices.
Overall functional wellness | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  Sheehan Disability Scale: a general self report in which participants indicate on a 11-point Likert scale ("Not at all" [0] - "Extremely" [10]) symptoms of disability and impairment have disrupted 3 general life categories work/school, social life, and family life/home responsibilities. Total score range for each category is 0-10, with higher ratings indicate a higher level of disruption in that life category.
Difficulties in performing life activities due to health conditions | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures World Health Organization Disability Assessment Schedule 2 (WHODAS 2.0): a 12-item self report questionnaire measuring the extent of difficulties experienced during specific life activities (ex. learning new tasks, getting dressed, maintaining friendships) from health conditions over the last 30 days on a 5-point Likert scale ("None" [0] - "Extreme/cannot do" [4]), and the estimated number of days in the last month that the individual felt impacted. Total score range 0-48, with higher scores representing higher degree of difficulty associated with health conditions.
Difficulties in performing work activities due to health conditions | From baseline to follow-up (immediate post intervention assessment)
  Outcome measures:
  Lam Employment Absence and Productivity Scale (LEAPS): A 7-item self report in which participants indicate on a 5-point Likert scale ("None of the time (0%)" [0] - "All of the time (100%)" [4]) the degree they have been bothered by issues impacting their work in the last 2 weeks (ex. productivity, energy, memory). Total score range is 0-28, with higher scores indicate higher degree of disruption in work tasks.
Workplace discrimination | From baseline to follow-up (immediate post intervention assessment)
  Outcome measure: The Workplace Gender Discrimination scale (6-item): Recruitment, promotions, pay, deployment, training and lay-offs. Respondents express degree of agreement on (4-point) Likert Scale [0]Strongly disagree to [3]Strongly agree. Total score is summed from 0 (strongly disagree) to 18 (strongly agree). 4 categories created: No gender discrimination in the workplace (scoring 0), low level (1-6), medium level (7-12), high level (13-18).
Gender-based workplace harassment | From baseline to follow-up (immediate post intervention assessment)
  Outcome measure: The Gender Experiences Questionnaire (GEQ) is a 20-item instrument that measures aspects of gender harassment in the workplace. Participants respond on a 5-point Likert scale: "Never" [1] to "Many Times" [5]. Total score range 20-100, higher scores indicate more frequent gender harassment.
Resting heart rate variability (HRV) | From baseline to follow-up (immediate post intervention assessment)
  Outcome Measures:
  Resting HRV will be computed from time and frequency domain parameters collected from the wearable HR monitors. Specifically, the time elapsed between two successive R-waves (i.e., heart beats) constitute an RR interval. The time difference between consecutive RR intervals are used to compute the root mean square of successive differences (RMSSD), which is used in the calculation of HRV in both high (HF) and low frequency (LF) domains. As such, calculation of RR intervals, RMSSD, and LF/HF ratios are in accordance with recommended standards of practice for HRV analysis. Increased HRV (msec) suggests improved vagal tone. We predict that resting HRV will significantly increase following completion of the AMT intervention.
Physiological recovery from acute stress | From baseline to follow-up (immediate post intervention assessment)
  Acute stress recovery will be assessed via a time domain measure of HRV (RMSSD), or the root mean square of successive differences between heart beats or RR intervals (in msec). A lower RMSSD indicates quicker physiological recovery from acute stress. We predict that recovery from acute stress will significantly improve following completion of the AMT intervention.
Respiratory Sinus Arrhythmia (RSA) | From baseline to follow-up (immediate post intervention assessment)
  Outcome Measures:
  RSA is operationalized by the degree of synchrony between HRV and respiratory frequency, both of which will be extracted from the raw data provided by the wearable HR monitor. Greater power at the respiratory frequency indicates a higher level of RSA and will be analyzed using the gold standard HRV analysis program, Kubios. We predict that RSA will significantly increase following completion of the AMT intervention.
Sex and gender differences in PTSI, occupational stress, and physiology | From baseline to follow-up (immediate post intervention assessment)
  Outcome Measures: All outcome measures listed above will be analyzed for differences according to self-reported sex and gender. Sex will be operationalized as self-reported biological sex assigned at birth and will include three possible responses: female, male, other. Gender will be operationalized as one of the following responses: female, male, non-binary, other, prefer not to disclose. Gender discrimination/ harassment will be explored as moderators of PTSI symptoms: We expect biological and gendered females to report more symptoms of PTSI, lower resilience at baseline, greater reduction of PTSI symptoms, greater increase in resilience at follow-up compared to biological and gendered males.

CONTACTS AND LOCATIONS:
Overall Officials: Judith P Andersen, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto Mississauga, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data (i.e., questionnaires, responses to intervention modules) will be transferred between members of the research team at University of Toronto (UofT) and other institutions in accordance with approved institutional data transfer agreements. Data from this study is confidential and participants' anonymity will be protected. Data from this research will be saved without mention of any participant names or other identifying information. All participants will be issued a unique identification number. A master file of the participant ID numbers and participant names will be maintained in a password-protected encrypted file at the PI's office at the University of Toronto and will be destroyed once the study has been completed. Participants will not be identified in any publication or reports and data. No data will be shared with the participant's employers, only aggregate study findings and de-identified results that are published in reports or publications.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Supporting information as listed above will become available after the study closure and publication of results (Anticipated 2025). Please check with the PI regarding further details
Access Criteria: contact PI

REFERENCES:
- [Derived] Andersen JP, Di Nota PM, Alavi N, Anderson G, Bennell C, McGregor C, Ricciardelli R, Scott SC, Shipley P, Vincent ML. A Biological Approach to Building Resilience and Wellness Capacity Among Police Exposed to Posttraumatic Stress Injuries: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 May 24;12:e33492. doi: 10.2196/33492. PMID 37223981